CLINICAL TRIAL: NCT04849819
Title: Effects of Systemic Diseases and Medications on Eye and Artificial Intelligence Model Development: a Multi-center Epidemiological Study
Brief Title: the SDMEAI Study: a Multi-center Epidemiological Study
Status: Not yet recruiting | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Haotian Lin, Vice President of Zhongshan Ophthalmic Center, Sun Yat-sen University
Other Study IDs: IIT2020023
Record Dates: First submitted 2021-04-15; First posted 2021-04-19 (Actual); Last update posted 2021-04-20 (Actual); Status verified 2021-04

CONDITIONS: Eye Involvement of Systemic Diseaes; Adverse Drug Effect on Eye; Artificial Intelligence
MeSH Terms: interventions — Adrenal Cortex Hormones; Biological Factors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- never receive systemic medications
- ever user of systemic medications
  Interventions: Drug: Corticosteroids, immunosuppressors, biological agents
- current user of systemic medications
  Interventions: Drug: Corticosteroids, immunosuppressors, biological agents

INTERVENTIONS:
Drug: Corticosteroids, immunosuppressors, biological agents — We do not prescribe new medications to patients but only observe their adverse effects on the eye.
  Groups: current user of systemic medications; ever user of systemic medications

SUMMARY:
A variety of diseases in the Department of Rheumatology, Immunology, Nephrology, and Gastroenterology can cause eye lesions, and medications can also bring various adverse reactions, which can seriously reduce the quality of patients' daily life, bring additional economic burdens, and even threaten the lives of patients. This study aims to recruit patients from the aboved-mentioned departments and conduct a cross-sectional and cohort study. On one hand, we plan to compare the epidemiological characteristics of ocular lesions of systemic diseases and eye adverse drug effects in patients with rheumatology, immunology, nephrology and gastroenterology, and summarized some epidemiological indices such as prevalence, high-risk factors, etc. On the other hand, we plan to develop an artificial intelligence model after collecting certain case data. By selecting risk factors related to the occurrence of ocular lesions, we aim to train models that can predict the ocular manifestations of systemic diseases and medications.

ELIGIBILITY:
Inclusion Criteria:

* Age 6-80 years old, gender is not limited
* patients who have been diagnosed with systemic diseases;
* patients who have ever or never used any ocular toxic drugs such as corticosteroids, chloroquine, etc.;
* no history of glaucoma, cataract, scleritis, uveitis, ocular trauma, etc. before enrollment;
* willing to complete follow-ups for at least 2 years.

Exclusion Criteria:

* Mainly use local therapies (intraocular, intra-articular and other non-systemic drug routes);
* history of intraocular surgery (such as lens implantation, vitrectomy, retinal photocoagulation);
* history of glaucoma, cataract, center serous retinopathy, etc.;
* history of various diseases (such as scleritis, uveitis, eye trauma, etc.) that may cause opacity of the eye under the posterior capsule;
* any other diseases or conditions that affect the observation, such as diabetes, low calcium convulsions, long-term exposure to radiation before enrollment;
* subjects with endogenous corticosteroids, or psychiatric diseases.

Ages: 6 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: We will recruit patients from the Sixth Affiliated Hospital, Sun Yat-Sen University and invite them to take ocular examinations in Zhongshan Ophthalmic Center, Sun Yat-Sen University. The Sixth Affiliated Hospital, Sun Yat-Sen University is a tertiary general hospital in Guangzhou, Guangdong, China. It has various departments, such as rheumatology and immunology department, nephrology departent and gastroenterology department, providing abundant cases of systemic diseases.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-04-22 (Estimated); Primary Completion 2025-04-22 (Estimated); Study Completion 2026-04-22 (Estimated)

PRIMARY OUTCOMES:
morbidity | 2021.4.22-2025.4.22
  Morbiditys of various ocular lesions.

CONTACTS AND LOCATIONS:
Overall Officials: Haotian Lin, Ph.D., Principal Investigator — Zhongshan Ophthalmic Center, Sun Yat-sen University

IPD SHARING:
Plan to Share IPD: Undecided